CLINICAL TRIAL: NCT04135794
Title: Magnetic Resonance-Guided Adaptive Radiotherapy (MRgART) Using an Integrated Magnetic Resonance Linear Accelerator (MRL)
Acronym: MRL1
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-5843
Record Dates: First submitted 2019-10-15; First posted 2019-10-23 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cancer
Keywords: MRL
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being done to help further understand how MR-guided adaptive RT in conjunction with the Integrated Magnetic Resonance Linear Accelerator (MRL) can improve patient outcomes. This study will include participants who will be receiving radiotherapy using the MRL machine to target their cancer more precisely. Participants will be asked to have a few extra MR scans taken during their RT planning and to complete a few quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with a diagnosis of cancer, regardless of clinical site or stage
* Planned to receive a course of MR-guided adaptive RT using the MRL
* Ability to provide informed consent

Exclusion Criteria:

* Patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cancer from any clinical site requiring radiotherapy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Local, regional and distant tumor control rates | Up to 5 years post-radiotherapy
  Refine our understanding of clinical scenarios where MRgART with the MRL improves patient outcomes and translate this new knowledge and new treatment approach to widespread clinical practice through the development and validation of efficient, cost-effective treatment processes.
Disease-free and overall survival rates | Up to 5 years post-radiotherapy
  Refine our understanding of clinical scenarios where MRgART with the MRL improves patient outcomes and translate this new knowledge and new treatment approach to widespread clinical practice through the development and validation of efficient, cost-effective treatment processes.
Complication rates measured using the Common Toxicity Criteria for Adverse Events | Within 3 months of completing treatment
  Refine our understanding of clinical scenarios where MRgART with the MRL improves patient outcomes and translate this new knowledge and new treatment approach to widespread clinical practice through the development and validation of efficient, cost-effective treatment processes.

SECONDARY OUTCOMES:
Patient experience and anxiety related to MR imaging and adaptive RT with the MR | Immediately after first MRL treatment visit
  Evaluate the patient experience during adaptive RT with the MRL using the Magnetic Resonance Imaging-Anxiety Questionnaire (MRI-AQ) which measures patient anxiety and tolerability of MR-related procedures
Patient experience and anxiety related to MR imaging and adaptive RT with the MR | Immediately after last MRL treatment visit
  Evaluate the patient experience during adaptive RT with the MRL using the EORTC satisfaction with cancer care core questionnaire (EORTC PATSAT-C33) and specific complementary outpatient module (EORTC OUT-PATSAT7)
Patient experience and anxiety related to MR imaging and adaptive RT with the MR | d prior to starting treatment with the MRL, immediately after the last MRL treatment, at the first follow-up visit and annually thereafter during follow-up (up to 5 years post treatment)
  Evaluate the patient experience during adaptive RT with the MRL using -The EORTC QLQ C30 quality of life questionnaire
Patient experience and anxiety related to MR imaging and adaptive RT with the MR | each ambulatory care and radiation treatment review clinic visit (up to 5 years post treatment)
  Evaluate the patient experience during adaptive RT with the MRL using complete the Edmonton Symptom Assessment Scale revised version (ESAS-r)

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada